CLINICAL TRIAL: NCT03031379
Title: Feasibility of Shortened Preoperative Fasts in Intubated ICU Patients Undergoing Tracheotomy
Brief Title: Shortened Preoperative Fasts in ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MMC-12-06-219
Record Dates: First submitted 2017-01-22; First posted 2017-01-25 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2012-02

CONDITIONS: Intubated ICU Patients

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A - control (No Intervention): standard fast, at least 6 hours prior to tracheotomy
- B - shortened fast (Experimental): fast of only 45 minutes prior to incision
  Interventions: Other: shortened fast

INTERVENTIONS:
Other: shortened fast — fast of 45 minutes prior to surgery as opposed to standard 6 hour fast
  Arms: B - shortened fast

SUMMARY:
Randomized controlled trial assessing the safety and benefits of shortening preoperative fasts on intubated ICU patients undergoing tracheotomy.

DETAILED DESCRIPTION:
Patients undergoing bedside tracheotomy in an ICU are enrolled and randomized into two groups. Arm A receive a standard fast of at least 6 hours. Arm B receive a shortened fast of only 45 minutes, just before the surgery begins. Patients will be monitored for aspiration, pneumonia and our ability to delivery better nutrition as a result of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* intubated ICU patient undergoing tracheotomy, receiving enteral nutrition, adult, proxy available for consent

Exclusion Criteria:

* pregnant, <18yo, cannot tolerate enteral feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Calories delivered | 72 hours
  Calories delivered before and after surgery

SECONDARY OUTCOMES:
Aspiration | 5 days
  intraoperative or postoperative aspiration

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States